CLINICAL TRIAL: NCT06007274
Title: Troponin to Detect Major Cardiovasculaire Advserse Events on Immune: a Case Control Retrospective Study
Brief Title: Troponin to Detect Major Cardiovasculaire Advserse Events on Immune Checkpoint Inhibitors
Acronym: TILT
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIO-04-2022
Record Dates: First submitted 2023-05-10; First posted 2023-08-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Immune Checkpoint Inhibitor; Cardiovascular Biomarkers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active surveillance by means of troponin measurements
  Interventions: Other: No intervention
- No active surveillance by means of troponin measurements

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: Active surveillance by means of troponin measurements

SUMMARY:
Recent guidelines suggest the use of troponin to detect immnune related cardiovascular advserse events in patients treated by immune checkpoint inhibitors for cancer.

However, there is no proof that patients on immune checkpoint inhibitors benefit from this active surveillance strategy. The suspicion of cardiovascular events may lead to the interruption of cancer therapies.

The TILT study aims at assessing: (i) the efficiency of troponin measurments in asymptomatic patients to prevent the further advent of major cardiovascular events; (ii) its safety in terms of cancer therapy completion.

DETAILED DESCRIPTION:
Retrospective two-center study comparing two groups of patients on immune checkpoint inhibitors:

* Group 1: active surveillance by serial troponin measures not prompted by cardiovascular symptoms ;
* Group 2: no troponin measures.

For any solid cancer or stage.

ELIGIBILITY:
Inclusion Criteria:

* All solid cancer patients treated by immune checkpoint inhibitors 2017-2022

Exclusion Criteria:

* Patients enrolled in an invterventional study (e.g., pharma trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult solid cancer patients receiving immune checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular event | 5 years
  Acute coronary syndrome, stroke, myocarditis, heart failure, sustained ventricular arrhymias, cardiovascular death

SECONDARY OUTCOMES:
Completion of cancer therapy as scheduled | 5 years
  Cardiovascular contre indication to immune checkpoint inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Mirabel, MD, PhD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided